CLINICAL TRIAL: NCT05259332
Title: Identification by Transcriptomic Approach of New Prognostic and Predictive Markers in a Cohort of Atypical Meningiomas and Immunohistochemical Applications
Brief Title: Identification by Transcriptomic Approach of New Prognostic and Predictive Markers in a Cohort of Atypical Meningiomas
Acronym: TransMenAtyp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Guillaume GAUCHOTTE, University professor and Hospital practitioner, Central Hospital, Nancy, France
Other Study IDs: 2020PI026
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Meningioma Atypical
Keywords: Transcriptome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor samples (atypical meningiomas WHO grade II)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determine by a transcriptomic approach new prognostic and predictive markers in atypical meningiomas (WHO grade II).

Retrospective observational study, on a cohort of 85 atypical meningiomas. Transcriptomic study first, on cryopreserved tumor samples. Then identify, thanks to the transcriptomic study, prognostic and predictive factors (study of the link between the quantity of certain RNA transcripts and progression-free survival). Finally, set up immunohistochemical applications, which can be used routinely by the pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Primary operated patients for an atypical meningioma (WHO grade II) in the Neurosurgery department of the University Hospital of Nancy.
* At least one postoperative follow-up visit.
* Adult patients (>18 yo) at the time of the intervention.
* Surgical excision.

Exclusion Criteria:

* History of meningioma in the same location.
* Neo-adjuvant treatment.
* Absence of non-objection form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the collection of biological samples from the Department of Pathological Anatomy and Cytology and the Biological Resource Center (CHRU Nancy).
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2022-02-25 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | through study completion an average of 5 years.
  Progression being defined by a growth (mm3) of the tumor objectified by imaging.

SECONDARY OUTCOMES:
Tumor volume assessed by imaging pre- and post-operative | before and within 3 months after surgery
  mm3; RECIST criteria
mRNA quantities of transcripts of interest | through study completion, an average of 1 year
  µg.mL-1
Radiotherapy-induced toxicity | within 5 years after radiotherapy
  CTCAE scale (Common Terminology Criteria for Adverse Events) v 4.0
Dose of corticosteroids before and after radiotherapy | within 6 months before and after radiotherapy
  in mg
Intra-observer, inter-observer and inter-laboratory intra-class correlation coefficients of immunohistochemical markers. | through study completion, an average of 1 year
  Kappa coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Guillaume GAUCHOTTE, Vandœuvre-lès-Nancy, Lorraine, France